CLINICAL TRIAL: NCT04850508
Title: Validation of the Advisor HD Grid Mapping Catheter in Atrial Fibrillation Ablation
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Vikas Kuriachan, Clinical Associate Professor (Cardiology/EP), University of Calgary
Other Study IDs: REB20-2140
Record Dates: First submitted 2021-04-13; First posted 2021-04-20 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Atrial Fibrillation
Keywords: Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mapping and ablation with the Advisor HD Grid catheter — After confirmation of isolation of the first pair of veins, the CMC-20 catheter will be exchanged for the HD Grid catheter. Using the HD Grid catheter, a new map of the left atrium will be made using the high-density settings. Together with the left atrium, the pulmonary veins will be mapped again in search of electro-anatomical gaps. Gaps are defined as a local area from the ablation line reaching inwards the pulmonary vein which still shows activation or fractionated potentials in line with atrial activation whilst pacing remote in the left atrium. The After mapping the first ablation side, the CMC-20 will be reinserted to repeat the protocol for the remaining pair of veins 30 minutes after ablation ended for that side.
  If gaps have been found, HD Grid guided additional ablation must be performed to achieve isolation in that vein until isolation is reconfirmed.

SUMMARY:
The primary study concept is to evaluate the superiority of the HD Grid high-density mapping catheter over the current standard 20-pole circular mapping catheter in pulmonary vein isolation (PVI) in atrial fibrillation. A minimum of 20 evaluable subjects with symptomatic atrial fibrillation scheduled for a clinically indicated first PVI ablation will be included.

DETAILED DESCRIPTION:
Background and Rationale:

The main target in atrial fibrillation ablation is the isolation of the pulmonary veins (PVI). This is performed by point-by-point ablation with radiofrequency energy creating 2 circles, one around the left superior and inferior pulmonary vein and one around the right superior and inferior pulmonary vein. The current standard of mapping the pulmonary vein ostia during PVI ablation is a 20-pole circumferential catheter (CMC-20) which collects anatomical and electrical information by moving it in the left atrium and making contact with the atrial wall. Isolation of pulmonary veins is confirmed by other methods such as bidirectional block across the ablation lesions.

New technological developments have resulted in high-density mapping, such as the Advisor HD Grid mapping catheter by Abbott. This catheter has a total of 16 electrodes configured in a 4 by 4 matrix. With each electrical wavefront being decomposed to 2 orthogonal vectors, every direction of a local wavefront should be detected by these configurations and thus overcoming the bipolar blindness.

Research Question and Objectives:

The primary objective of this study is to demonstrate the superiority of the HD Grid catheter when compared to the CMC-20 catheter in atrial fibrillation ablation.

The primary endpoint is the mean number of gaps identified per patient, and their location identified by the HD Grid catheter after standard PVI procedure with the CMC-20 catheter.

Secondary endpoints are:

* A per vein analysis will be performed for the presence of gaps and for the mean number of gaps.
* A per pair of veins (left and right separately) analysis will be performed for the presence of gaps and for the mean number of gaps.
* Left atrial mapping time for both the CMC-20 and the HD Grid catheter
* Discrepancies in the prevalence of low voltage areas defined as a voltage <0.50 mV between the CMC-20 and HD Grid catheter in sinus rhythm.

Design:

Prospective, single arm, single center, superiority study with comparison of standard 20-pole circular mapping catheter and the new HD Grid multipolar catheter.

A minimum of 20 evaluable subjects with drug refractory, symptomatic atrial fibrillation scheduled for first PVI ablation will be enrolled over a period of 12 months.

Data collection:

Demographic, clinical and AF-related information will be collected prior to the procedure. Procedure related information will be collected directly after the procedure. All data will be collected in RedCap.

Procedure:

First, a standard PVI procedure is performed. After completion of the ablation lesions, isolation of the pulmonary veins will be confirmed using the standard CMC-20 catheter. If isolation is confirmed, the CMC-20 catheter will be exchanged for the HD Grid catheter. Using the HD Grid catheter, a new map of the left atrium will be made using the high-density settings. Together with the left atrium, the pulmonary veins will be mapped again in search of electro-anatomical gaps. Gaps are defined as a local area from the ablation line reaching inwards the pulmonary vein which still shows activation or fractionated potentials in line with atrial activation whilst pacing remote in the left atrium. The prevalence and location of these gaps will be collected using the map. If gaps have been found, HD Grid guided additional ablation must be performed to achieve isolation in that vein.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic paroxysmal or persistent atrial Fibrillation.1
2. Patients referred for a clinically indicated catheter ablation with a plan for PVI only.
3. 18-85 year of age at time of consent.
4. Able and willing to comply with all protocol requirements.
5. Signed patient Informed Consent (ICF).

Exclusion Criteria:

1. History of prior left-sided catheter or surgical ablation for AF or atypical atrial flutter, including MAZE or mini MAZE. Prior ablation for typical atrial flutter or left-sided ablation for WPW, AV-node reentry tachycardia or right-sided focal ectopic atrial tachycardia may be included.
2. Planned for left atrial ablation beyond PVI.
3. Uncontrolled heart Failure or NYHA Class III or IV heart failure.
4. Left ventricular ejection fraction < 35 %
5. Left atrial size > 55 mm diameter on echocardiogram.
6. Severe Pulmonary Hypertension
7. Reversible causes of AF (electrolyte imbalance, thyroid disease…)
8. Poor candidate for general anesthesia or deep sedation
9. Anticipated survival < 1 year
10. MI or CABG within 3 months, severe valvular disease
11. Any documented thromboembolic event within 6 months.
12. Contraindication to systemic oral anticoagulation therapy.
13. Significant congenital anomaly or medical condition that may affect the integrity of study data.
14. Women who are pregnant or breastfeeding.
15. Active enrollment in another investigational study involving a drug or device.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with drug refractory, symptomatic atrial fibrillation scheduled for first PVI ablation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Number of gaps | During the ablation procedure.
  The primary endpoint is the mean number of gaps identified per patient identified by the HD Grid catheter after standard PVI procedure with the CMC-20 catheter.
Location of gaps | During the ablation procedure.
  The co-primary endpoint is the location of the gaps identified per patient by the HD Grid catheter after standard PVI procedure with the CMC-20 catheter.

SECONDARY OUTCOMES:
Per vein analysis for the presence of any gap. | During the ablation procedure.
  A per vein analysis will be performed for the presence of any gap as a binary outcome.
Per vein analysis for the mean number of gaps. | During the ablation procedure.
  A per vein analysis will be performed for the mean number of gaps.
Per pair of veins analysis for the presence of any gap. | During the ablation procedure.
  A per pair of veins (left and right separately) analysis will be performed for the presence of any gap as a binary outcome.
Per pair of veins analysis for the mean number of gaps. | During the ablation procedure.
  A per pair of veins (left and right separately) analysis will be performed for the mean number of gaps.
Mapping time | During the ablation procedure.
  Left atrial mapping time for both the CMC-20 and the HD Grid catheter
Discrepancies | During the ablation procedure.
  Discrepancies in the prevalence of low voltage areas defined as a voltage <0.50 mV between the CMC-20 and HD Grid catheter in sinus rhythm.

CONTACTS AND LOCATIONS:
Overall Officials: Vikas P Kuriachan, MD, Principal Investigator — Libin Cardiovascular Institute of Alberta, University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Given the small number of patients in the study individual treatments and outcomes maybe looked at.

REFERENCES:
- [Background] Porterfield C, J Gora P, Wystrach A, Rossi P, Rillo M, A Sebag F, Giuggia M, Mantica M, Dorszewski A, Eldadah Z, Volpicelli M, Bottoni N, Jons C, T Hollis Z, Dekker L, Mathew S, Schmitt J, Nilsson K. Confirmation of Pulmonary Vein Isolation with High-Density Mapping: Comparison to Traditional Workflows. J Atr Fibrillation. 2020 Apr 30;12(6):2361. doi: 10.4022/jafib.2361. eCollection 2020 Apr-May. PMID 33024494
- [Derived] Vandenberk B, Quinn FR, Barmby J, Wilton SB, Kuriachan V. High-density mapping improves detection of conduction gaps after pulmonary vein isolation ablation with a circular mapping catheter. J Interv Card Electrophysiol. 2023 Sep;66(6):1401-1410. doi: 10.1007/s10840-022-01434-3. Epub 2022 Dec 3. PMID 36462064